CLINICAL TRIAL: NCT03381248
Title: A Prospective, Multi-center, Randomized, Clinical Trial Evaluating the Safety and Effectiveness of Using COOLIEF™ Cooled Radiofrequency Probe to Create Lesions of the Genicular Nerves and Comparing a Single Injection of Hyaluronic Acid in the Management of Knee Pain
Brief Title: Cooled Radiofrequency vs. Hyaluronic Acid to Manage Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avanos Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105-17-0001
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Results first posted 2020-05-22 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis of the Knee
Keywords: randomized clinical trial; osteoarthritis; radiofrequency ablation; knee; genicular; cross-over; viscosupplementation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Hyaluronic Acid; Viscosupplementation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cooled Radiofrequency (Experimental): Cooled radiofrequency energy will be delivered to study subjects' knees to ablate culprit sensory nerves and reduce knee pain. Subjects in this group will be followed for 12 months post-procedure.
  Interventions: Device: Cooled Radiofrequency
- Hyaluronic Acid, then Cooled Radiofrequency (Active Comparator): Hyaluronic acid injections will be administered to study subjects' knees to reduce knee pain. Subjects in this group will have the option to crossover to receive cooled radiofrequency after 6-months. Crossover subjects will be followed for an additional 6 months post-procedure. Non-crossover subjects will continue to be followed until the 12-month timepoint.
  Interventions: Other: Hyaluronic Acid Injection; Other: Crossover from Hyaluronic Acid Injection to Cooled Radiofrequency

INTERVENTIONS:
Device: Cooled Radiofrequency — Delivery of energy to ablate sensory nerves via cooled radiofrequency probe.
  Other Names: Coolief
  Arms: Cooled Radiofrequency
Other: Hyaluronic Acid Injection — Delivery of hyaluronic acid into knee by injection with needle to reduce knee pain.
  Other Names: Viscosupplementation
  Arms: Hyaluronic Acid, then Cooled Radiofrequency
Other: Crossover from Hyaluronic Acid Injection to Cooled Radiofrequency — Delivery of hyaluronic acid into knee by injection with needle to reduce knee pain. After 6 months, qualifying subjects in this group will have the option to crossover to receive cooled radiofrequency treatment.
  Other Names: Viscosupplementation; Cooled Radiofrequency
  Arms: Hyaluronic Acid, then Cooled Radiofrequency

SUMMARY:
This is a prospective, randomized, multicenter comparison study examining the outcomes of subjects with osteoarthritis and knee pain undergoing a procedure to create a radiofrequency lesion of the genicular nerves with the Cooled Radiofrequency Ablation (CRFA) system compared to subjects receiving Hyaluronic Acid (HA). Approximately 168 subjects will be enrolled into this study, with subjects undergoing either CRFA or HA injection in a 1:1 randomization scheme. Follow-up will be conducted for 12 months post-CRFA, with the primary endpoint being completed at month 6. Subjects randomized to the comparison (HA) group will have the option to cross-over to the neurotomy group after completing the 6-month endpoint assessment. They will be followed for an additional 6 months. Pain, overall outcome, quality of life, pain medication use, and adverse events will be compared between the two treatment groups to determine success. Subjects who were randomized to and received COOLIEF* as their initial treatment will have the option to add 2 additional visits at 6-month intervals, representing 18 and 24 months post initial treatment.

DETAILED DESCRIPTION:
The COOLIEF™ system components utilized in the study are the same in form and function regardless of specific product branding (COOLIEF* or SInergy*). The COOLIEF™ system is comprised of three primary components (collectively known as 'disposables') and is used in conjunction with the Pain Management generator, pump unit, connector cables (collectively known as 'Hardware') and dispersive electrodes (also known as 'grounding pads'):

* Cooled Radiofrequency Sterile Tube Kit (sterile, single use, non-body contact): It is used for closed-loop circulation of sterile water through a Halyard Health* Cooled Radiofrequency Probe. It includes a burette and tubing.
* Cooled Radiofrequency Introducer (sterile, single use): It is to be used with the Probes only. The Cooled Radiofrequency Introducer provides a path for the Probe to the targeted nervous tissue.
* Cooled Radiofrequency Probe (sterile, single use): It is inserted through an Introducer into or near nervous tissue. The active tip extends 4mm from the introducer and delivers energy. Sterile water circulates internally to cool the Probe while it delivers radiofrequency energy. A thermocouple in the Probe measures the cooled electrode temperature throughout the procedure.

The product is comprised of an electrically insulated shaft with an active tip that functions as an electrode for radiofrequency energy delivery, a handle, tubes with luer locks and a cable with a 7-pin connector. The Introducer includes an insulated stainless steel cannula and a stylet. The Tube Kit is comprised of a burette and flexible tubing fitted with luer locks for connection to the Probe. The Probe, Introducer, and Tube Kit are ethylene oxide sterilized and supplied sterile. These components can be packaged together in a kit or as separate components. The devices should be stored in a cool, dry environment. The Instructions For Use (IFU) documents (Appendix 1) are included in each kit.

Halyard Health maintains a list of all model numbers and sizes for the system components.

The control product/device, Synvisc-One® (hylan G-F 20) (HA), is an elastoviscous high molecular weight fluid containing hylan A and hylan B polymers produced from chicken combs. Hylans are derivatives of hyaluronan (sodium hyaluronate). Hylan G-F 20 is unique in that the hyaluronan is chemically crosslinked. Hyaluronan is a long-chain polymer containing repeating disaccharide units of Na-glucuronate-N-acetylglucosamine.

Synvisc-One is a single injection regimen therapy indicated for the treatment of pain in Osteoarthritis of the knee in patients who have failed to respond adequately to conservative nonpharmacologic therapy and simple analgesics, e.g., acetaminophen.

Following treatment, subjects in the CRF treatment group will follow up at 1, 3, 6 and 12 months. These subjects will then have the option to return for two additional visits at 18 and 24 months. Subjects initially randomized to the comparison (HA) group will follow up at 1, 3, and 6 months, and then be given the option to receive crossover CRF treatment. If crossover CRF treatment was received, subjects will return for follow up visits at 1, 3, and 6 months post-treatment. If crossover treatment was not received, subjects will return for their final 12 month visit.

Study Duration:

* Treatment Group: Up to 24 months following index procedure
* Control Group: Up to 13 months, depending upon receipt of cross-over procedure.

Effectiveness Endpoints:

* Numeric Rating Scale (NRS, Usual Level of Pain)
* Western Ontario & McMaster University Osteoarthritis Index (WOMAC)
* EQ-5D-5L Health-Related Quality of Life Questionnaire
* Global Perceived Effect Scale

ELIGIBILITY:
INCLUSION CRITERIA

1. Age ≥ 21 years
2. Able to understand the informed consent form and provide written informed consent and able to complete outcome measures
3. Chronic knee pain for longer than 6 months that interferes with functional activities (for example, ambulation, prolonged standing, etc.)
4. Continued pain in the target knee despite at least 3 months of conservative treatments, including activity modification, home exercise, protective weight bearing, and/or analgesics (for example, acetaminophen or non-steroidal anti-inflammatory drugs [NSAIDs])
5. Positive response (defined as a decrease in numeric pain scores of at least 50%) to a single genicular nerve block of the index knee
6. Pain on NRS ≥ 6 on an 11-point scale for the index knee
7. Radiologic confirmation of arthritis (x-ray/MRI/CT) of Osteoarthritis (OA) grade of 2 (mild), 3 (moderate) or 4 (severe) noted within 6 months for the index knee
8. An intra-articular hyaluronic acid injection is indicated as an appropriate treatment option
9. WOMAC Knee Score group at baseline of Score of ≥ 2 (0 to 4 scale) on WOMAC question 1 (Pain) and a mean score of ≥ 1.5 on all five questions of the WOMAC pain subscale.
10. Analgesics including membrane stabilizers such as Neurontin/gabapentin and antidepressants for pain such as Cymbalta/duloxetine must be clinically stable (defined as stable dosage for ≥ 6 weeks prior to the screening visit) and shall not change during the course of the study without approval of the investigator
11. Agree to see one physician (study physician) for knee pain during the study period
12. Willing to utilize double barrier contraceptive method if of child bearing potential.
13. Willing to delay any surgical intervention for the index knee for the period of the study follow up
14. Willingness to provide informed consent and to comply with the requirements of this protocol for the full duration of the study

EXCLUSION CRITERIA

1. Evidence of inflammatory arthritis (for example, rheumatoid arthritis) or other systemic inflammatory condition (for example, gout, fibromyalgia) that could cause knee pain
2. Evidence of neuropathic pain affecting the index knee
3. Previous or pending lower limb amputation
4. Intra-articular steroid injection into the index knee within 90 days from randomization
5. Hyaluronic acid injection, platelet rich plasma (PRP), stem cell, or arthroscopic debridement/lavage injection into the index knee within 180 days from randomization
6. Prior radiofrequency ablation of the genicular nerves of the index knee
7. Prior partial, resurfacing, or total knee arthroplasty of the index knee (residual hardware)
8. Clinically significant ligamentous laxity of the index knee
9. Clinically significant valgus/varus deformities or evidence of pathology (other than osteoarthritis of knee) that materially affects gait or function of the knee or is the underlying cause of the knee pain and/or functional limitations
10. Body mass index (BMI) > 40 kg/m2
11. Extremely thin patients and those with minimal subcutaneous tissue thickness that would not accommodate a radiofrequency lesion of up to 14 mm in diameter to limit the risk of skin burns
12. Pending or active compensation claim, litigation or disability remuneration (secondary gain)
13. Pregnant, nursing or intent on becoming pregnant during the study period
14. Chronic pain associated with significant psychosocial dysfunction
15. Beck's Depression Index score of > 22 (indicates clinically depressed state)
16. Allergies to any of the medications to be used during the procedures, including known hypersensitivity (allergy) to hyaluronate preparations or allergies to avian or avian-derived products (including eggs, feathers, or poultry)
17. Active joint infection or systemic or localized infection at needle entry sites (subject may be considered for inclusion once infection is resolved)
18. History of uncontrolled coagulopathy, ongoing coagulation treatment that cannot be safely interrupted for procedure, or unexplained or uncontrollable bleeding that is uncorrectable.
19. Identifiable anatomical variability that would materially alter the procedure as described in the protocol
20. Within the preceding 2 years, subject has suffered from active narcotic addiction, substance, or alcohol abuse
21. Current prescribed opioid medications greater than 60 morphine equivalent daily opioid dose
22. Uncontrolled immunosuppression (e.g. AIDS, cancer, diabetes, etc.)
23. Subject currently implanted with pacemaker, stimulator or defibrillator.
24. Participating in another clinical trial/investigation within 30 days prior to signing informed consent
25. Subject unwilling or unable to comply with follow up schedule or protocol requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia F Chen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (10):
- United States (10):
  - Lyman Medical Research, Coeur d'Alene, Idaho
  - Ocshner Baptist Clinical Trials Unit, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - University Orthopedics Center, Altoona, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Piedmont Comprehensive Pain Management, Anderson, South Carolina
  - University of Virginia, Charlottesville, Virginia
  - Virginia iSpine Physicians, Richmond, Virginia

REFERENCES:
- [Derived] Chen AF, Khalouf F, Zora K, DePalma M, Kohan L, Guirguis M, Beall D, Loudermilk E, Pingree MJ, Badiola I, Lyman J. Cooled radiofrequency ablation provides extended clinical utility in the management of knee osteoarthritis: 12-month results from a prospective, multi-center, randomized, cross-over trial comparing cooled radiofrequency ablation to a single hyaluronic acid injection. BMC Musculoskelet Disord. 2020 Jun 9;21(1):363. doi: 10.1186/s12891-020-03380-5. PMID 32517739

RESULTS

PARTICIPANT FLOW:
Groups:
- Cooled Radiofrequency: Cooled radiofrequency energy will be delivered to study subjects' knees to ablate culprit sensory nerves and reduce knee pain
  Cooled Radiofrequency: Delivery of energy to ablate sensory nerves via cooled radiofrequency probe
- Hyaluronic Acid Injection, Then Cooled Radiofrequency Crossover Option: Hyaluronic acid injections will be administered to study subjects' knees to reduce knee pain. Qualifying study subjects will then have the option to crossover to receive CRFA at 3 months.
  Hyaluronic Acid: Delivery of hyaluronic acid into knee by injection with needle to reduce knee pain
  Cooled Radiofrequency: Delivery of energy to ablate sensory nerves via cooled radiofrequency probe
Period: 0-6 Months
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection, Then Cooled Radiofrequency Crossover Option
Started | 89 | 88
Completed (Completion is with respect to the 6-month primary outcome.) | 76 | 82
Not Completed | 13 | 6
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Planning another procedure | 1 | 2
Period: 6-12 Months
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection, Then Cooled Radiofrequency Crossover Option
Started | 76 | 82
Received Crossover Treatment | 0 | 68
Completed | 66 | 73
Not Completed | 10 | 9
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Planning another procedure | 6 | 2
Period: 12 - 24 Months (Extension Study)
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection, Then Cooled Radiofrequency Crossover Option
Started | 36 (9 subjects ineligible as site was not participating in extension phase of study; 21 additional eligible subjects chose not to participate in extension phase of study) | 0
Completed | 27 | 0
Not Completed | 9 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Received another procedure | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hyaluronic Acid Injection: Hyaluronic acid injections will be administered to study subjects' knees to reduce knee pain
  Hyaluronic Acid: Delivery of hyaluronic acid into knee by injection with needle to reduce knee pain
- Total: Total of all reporting groups
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection | Total
Number analyzed (Participants) | 89 | 88 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.7) | 63.1 (9.7) | 63.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 106
  Male | 37 | 34 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 8 | 11
  White | 83 | 80 | 163
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 89 | 88 | 177

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS)
Description: The proportion of subjects whose knee pain is reduced by ≥ 50% based on the NRS. The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals the "worst pain". There are no sub-scales.
Time Frame: Baseline to 6 month study visit
Population: 76 of the 89 originally-randomized study subjects in the Cooled Radiofrequency group completed this 6-month outcome. 82 of the originally-randomized 88 study subjects in the Hyaluronic Acid Injection group completed this 6-month outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection, Then Cooled Radiofrequency Crossover Option
Number analyzed (Participants) | 76 | 82
Participants | 54 | 31

2. Primary Outcome: Safety: The Proportion of Subjects Experiencing Adverse Events Through Final Follow up.
Description: Safety: The proportion of subjects experiencing adverse events through final follow up.
Time Frame: Baseline to 12 month study visit
Measure: Count of Participants; unit: Participants
Groups:
- Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency: Subjects initially randomized to the Control (Hyaluronic Acid) group who remained in significant pain at 6 months who chose to receive crossover Cooled Radiofrequency treatment.
  Hyaluronic Acid: Delivery of hyaluronic acid into knee by injection with needle to reduce knee pain
  Cooled Radiofrequency: Delivery of energy to ablate sensory nerves via cooled radiofrequency probe
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection | Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency
Number analyzed (Participants) | 89 | 88 | 68
Participants | 78 | 48 | 38

3. Secondary Outcome: Numeric Rating Scale
Description: The proportion of subjects whose knee pain is reduced from baseline by ≥ 50% based on the NRS. The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals the "worst pain". There are no sub-scales.
Time Frame: Baseline (or date of crossover for Crossover group subjects) to 12 month study visit
Population: 66 of the 89 originally-randomized study subjects in the Cooled Radiofrequency group completed this 12-month outcome measure. 62 of the originally-randomized 88 study subjects in the Hyaluronic Acid Injection group chose to crossover to receive Cooled Radiofrequency treatment and completed this 12-month outcome. 11 of the originally-randomized subjects in this group who elected not to crossover completed this 12-month outcome.
Measure: Count of Participants; unit: Participants
Groups:
- CROSSOVER From Hyaluronic Acid Injection to Cooled Radiofrequency: Subjects initially randomized to the Control (Hyaluronic Acid) group who remained in significant pain at 6 months who chose to receive crossover Cooled Radiofrequency treatment.
  Cooled radiofrequency energy will be delivered to study subjects' knees to ablate culprit sensory nerves and reduce knee pain
  Cooled Radiofrequency: Delivery of energy to ablate sensory nerves via cooled radiofrequency probe
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection | CROSSOVER From Hyaluronic Acid Injection to Cooled Radiofrequency
Number analyzed (Participants) | 66 | 11 | 62
Participants | 43 | 10 | 40

4. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The change in WOMAC score from baseline to 6 months. This outcome instrument is composed of three sub-scales, including "Pain" (5 questions), "Stiffness" (2 questions), and "Physical Function" (17 questions). The point range for each sub-scale question is from 0 to 4, with "0" indicating the best study subject condition and "4" indicating the worst study subject condition. Thus, the minimum score per sub-scale is 0, and the maximum is 20, 8, and 68 for "Pain", Stiffness", and "Physical Function", respectively. The minimum and maximum possible scores for the entire instrument are 0 (best study subject condition) and 96 (worst study subject condition).
Time Frame: Baseline to 6 month study visit
Population: The 'change from baseline' was unable to be calculated for one of the CRFA-randomized subjects as appropriate baseline measurements for this outcome measure were not collected. The comparison could not be performed for this subject. Therefore, the Overall Number of Participants Analyzed in this group is reduced by one.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection
Number analyzed (Participants) | 75 | 82
units on a scale | 31.5 (23.0) | 14.8 (19.4)

5. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The change in WOMAC score from baseline to 12 months. This outcome instrument is composed of three sub-scales, including "Pain" (5 questions), "Stiffness" (2 questions), and "Physical Function" (17 questions). The point range for each sub-scale question is from 0 to 4, with "0" indicating the best study subject condition and "4" indicating the worst study subject condition. Thus, the minimum score per sub-scale is 0, and the maximum is 20, 8, and 68 for "Pain", Stiffness", and "Physical Function", respectively. The minimum and maximum possible scores for the entire instrument are 0 (best study subject condition) and 96 (worst study subject condition).
Time Frame: Baseline (or date of crossover for Crossover group subjects) to 12 month study visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency: Subjects initially randomized to the Control (Hyaluronic Acid) group who remained in significant pain at 6months who chose to receive crossover Cooled Radiofrequency treatment.
  Cooled radiofrequency energy will be delivered to study subjects' knees to ablate culprit sensory nerves and reduce knee pain
  Cooled Radiofrequency: Delivery of energy to ablate sensory nerves via cooled radiofrequency probe
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection | Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency
Number analyzed (Participants) | 65 | 11 | 62
units on a scale | 30.7 (25.2) | 32.1 (18.3) | 18.1 (22.1)

6. Other Pre Specified Outcome: EQ-5D-5L
Description: The change in measured EQ-5D-5L scale from baseline to 6 months. This outcome instrument is composed of five sub-scales containing five questions each. The point range for each sub-scale is from 1 to 5, with "1" indicating the best study subject condition and "5" indicating the worst study subject condition. Thus, the minimum and maximum scores per sub-scale are 1 and 5, respectively, and such scores for the entire instrument are 5 (best study subject condition) and 25 (worst study subject condition). The sub-scale topics are: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression.
Time Frame: Baseline to 6 month study visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection
Number analyzed (Participants) | 75 | 82
units on a scale | 0.12 (0.14) | 0.06 (0.15)

7. Other Pre Specified Outcome: EQ-5D-5L
Description: The change in measured EQ-5D-5L scale from baseline to 12 months. This outcome instrument is composed of five sub-scales containing five questions each. The point range for each sub-scale is from 1 to 5, with "1" indicating the best study subject condition and "5" indicating the worst study subject condition. Thus, the minimum and maximum scores per sub-scale are 1 and 5, respectively, and such scores for the entire instrument are 5 (best study subject condition) and 25 (worst study subject condition). The sub-scale topics are: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression.
Time Frame: Baseline (or date of crossover for Crossover group subjects) to 12 month study visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection | Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency
Number analyzed (Participants) | 65 | 11 | 62
units on a scale | 0.12 (0.14) | 0.14 (0.14) | 0.08 (0.15)

8. Other Pre Specified Outcome: Global Perceived Effect
Description: Number of participants with improvement measured by the Global Perceived Effect scale. The Global Perceived Effect is a 7-point scale: 1 point = "worst ever", 2 points = "much worse", 3 points = "worse", 4 points = "not improved but not worse", 5 points = "improved", 6 points = "much improved", 7 points = "best ever". There are no sub-scales. Number of participants scoring at either 5, 6, or 7 points on the Global Perceived Effect scale are reported.
Time Frame: Baseline to 6 month study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection
Number analyzed (Participants) | 76 | 82
Participants | 55 | 33

9. Other Pre Specified Outcome: Global Perceived Effect
Description: as for outcome 8
Time Frame: Baseline (or date of crossover for Crossover group subjects) to 12 month study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection | Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency
Number analyzed (Participants) | 66 | 11 | 62
Participants | 42 | 8 | 39

10. Other Pre Specified Outcome: Numeric Rating Scale
Description: as for outcome 3
Time Frame: Baseline to 18 month study visit
Population: 32 of the 36 study subjects who elected to participate in the CRFA extension phase of the study completed this 18-month outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 32
Participants | 22

11. Other Pre Specified Outcome: Numeric Rating Scale
Description: as for outcome 3
Time Frame: Baseline to 24 month study visit
Population: 27 of the 36 study subjects who elected to participate in the CRFA extension phase of the study completed this 24-month outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 27
Participants | 17

12. Other Pre Specified Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The change in WOMAC score from baseline to 18 months. This outcome instrument is composed of three sub-scales, including "Pain" (5 questions), "Stiffness" (2 questions), and "Physical Function" (17 questions). The point range for each sub-scale question is from 0 to 4, with "0" indicating the best study subject condition and "4" indicating the worst study subject condition. Thus, the minimum score per sub-scale is 0, and the maximum is 20, 8, and 68 for "Pain", Stiffness", and "Physical Function", respectively. The minimum and maximum possible scores for the entire instrument are 0 (best study subject condition) and 96 (worst study subject condition).
Time Frame: Baseline to 18 month study visit
Population: Extension study subjects with 18-month data available for analysis for this outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 30
units on a scale | 29.3 (25.3)

13. Other Pre Specified Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The change in WOMAC score from baseline to 24 months. This outcome instrument is composed of three sub-scales, including "Pain" (5 questions), "Stiffness" (2 questions), and "Physical Function" (17 questions). The point range for each sub-scale question is from 0 to 4, with "0" indicating the best study subject condition and "4" indicating the worst study subject condition. Thus, the minimum score per sub-scale is 0, and the maximum is 20, 8, and 68 for "Pain", Stiffness", and "Physical Function", respectively. The minimum and maximum possible scores for the entire instrument are 0 (best study subject condition) and 96 (worst study subject condition).
Time Frame: Baseline to 24 month study visit
Population: Extension study subjects with 24-month data available for analysis for this outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 26
units on a scale | 41.3 (29.9)

14. Other Pre Specified Outcome: EQ-5D-5L
Description: The change in measured EQ-5D-5L scale from baseline to 18 months. This outcome instrument is composed of five sub-scales containing five questions each. The point range for each sub-scale is from 1 to 5, with "1" indicating the best study subject condition and "5" indicating the worst study subject condition. Thus, the minimum and maximum scores per sub-scale are 1 and 5, respectively, and such scores for the entire instrument are 5 (best study subject condition) and 25 (worst study subject condition). The sub-scale topics are: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression.
Time Frame: Baseline to 18 month study visit
Population: Extension study subjects with 18-month data available for analysis for this outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 30
units on a scale | 0.15 (0.14)

15. Other Pre Specified Outcome: EQ-5D-5L
Description: The change in measured EQ-5D-5L scale from baseline to 24 months. This outcome instrument is composed of five sub-scales containing five questions each. The point range for each sub-scale is from 1 to 5, with "1" indicating the best study subject condition and "5" indicating the worst study subject condition. Thus, the minimum and maximum scores per sub-scale are 1 and 5, respectively, and such scores for the entire instrument are 5 (best study subject condition) and 25 (worst study subject condition). The sub-scale topics are: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression.
Time Frame: Baseline to 24 month study visit
Population: Extension study subjects with 18-month data available for analysis for this outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 26
units on a scale | 0.07 (0.14)

16. Other Pre Specified Outcome: Global Perceived Effect
Description: as for outcome 8
Time Frame: Baseline to 18 month study visit
Population: Extension study subjects with 18-month data available for analysis for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 32
Participants | 24

17. Other Pre Specified Outcome: Global Perceived Effect
Description: as for outcome 8
Time Frame: Baseline to 24 month study visit
Population: Extension study subjects with 18-month data available for analysis for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 27
Participants | 17

18. Other Pre Specified Outcome: Safety: The Proportion of Subjects Experiencing Adverse Events Between 12 - 24 Months (Extension)
Description: Safety: The proportion of subjects experiencing adverse events between 12 - 24 months (Extension)
Time Frame: 12 month study visit to 24 month study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency
Number analyzed (Participants) | 36
Participants | 19

ADVERSE EVENTS:
Time Frame: Total Study: Baseline to 24 months
Description: CRFA group includes all AEs from subjects randomized to and treated with Cooled Radiofrequency Ablation (from baseline to 24 months, including extension). HA group includes all AEs from subjects randomized to and treated with Hyaluronic Acid Injections (from baseline to 6 months) and AEs from subjects who did not receive crossover CRFA treatment (from 6 to 12 months). Crossover group includes all AEs experienced by HA subjects following receipt of crossover CRFA treatment (from 6 to 12 months).
Arm/Group | Cooled Radiofrequency | Hyaluronic Acid Injection | Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/88 | 0/68
Serious Adverse Events (participants affected / at risk) | 13/89 | 2/88 | 1/68
Other Adverse Events (participants affected / at risk) | 85/89 | 46/88 | 37/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooled Radiofrequency (N=89) | Hyaluronic Acid Injection (N=88) | Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency (N=68)
Cardiovascular (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0)
Genitourinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
H.E.E.N.T (General disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) — (Procedure)
Neurological (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Other (General disorders) | 1 (1) | 0 (0) | 0 (0) — (Fall)
Blood/Lymphatic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Endocrine/Metabolic (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0)
Extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooled Radiofrequency (N=89) | Hyaluronic Acid Injection (N=88) | Crossover From Hyaluronic Acid Injection to Cooled Radiofrequency (N=68)
Blood/Lymphatic/Infection (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Cardiovascular (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
Endocrine/Metabolic (Endocrine disorders) | 4 (4) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Genitourinary (Renal and urinary disorders) | 1 (1) | 2 (6) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 83 (127) | 38 (49) | 29 (50)
Neurological (Nervous system disorders) | 8 (8) | 2 (2) | 3 (3)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 1 (1)
Other (General disorders) | 13 (16) | 10 (11) | 9 (10)
H.E.E.N.T / Infection (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03381248/Prot_SAP_000.pdf